CLINICAL TRIAL: NCT06563362
Title: Personalized Volume-deescalated Elective Nodal Irradiation in Oropharyngeal Head and Neck
Brief Title: Personalized Volume-deescalated Elective Nodal Irradiation in Oropharyngeal Head and Neck Squamous Cell Carcinoma
Acronym: DeEscO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other); Ospedale Regionale Bellinzona e Valli (Other); Réseau Hospitalier Neuchâtelois (Other); Kantonsspital Aarau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DeEscO
Record Dates: First submitted 2024-08-08; First posted 2024-08-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Oropharynx Cancer
Keywords: head and neck cancer; radiotherapy; elective CTV; clinical target volume; de-escalation
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elective target volume de-escalation arm (Experimental): Target volume de-escalation
  Interventions: Radiation: De-escalation of irradiated volume

INTERVENTIONS:
Radiation: De-escalation of irradiated volume — De-escalation of elective clinical target volumes as recommended by a model-based approach

SUMMARY:
Multicentric prospective model-based de-escalation of the elective clinical target volumes (CTV) in radiotherapy of oropharyngeal carcinoma of all stages with the goal to reduce toxicity.

The study investigates the feasibility of this approach as measured by the number of expected out-of-field recurrencies based on the individual patient's state of disease progression and risk factors

DETAILED DESCRIPTION:
Local treatment of squamous cell carcinoma (SCC) of the oropharynx can consist of surgery, radiotherapy, or a combination of both. When treated with radiation, the target volume contains not only the primary tumor and clinically detected lymph node metastases. In addition, a large part of the lymph drainage system of the neck which is at risk of harboring occult metastases is irradiated, the so called "elective clinical target volume (CTV)". This elective CTV is currently based on clinical recommendations, but there is limited data and evidence on (occult) lymphatic spread and the required size of the elective CTV. This standard radiotherapy approach is associated with early and late toxicity. Toxicities such as pain, dermatitis, mucositis, but also long-term sequela like swallowing dysfunction, lymphedema and dysgeusia are commonly described, which can even lead to hospitalization or long-term symptoms with subsequent life-quality impairment.

A de-escalation of the treatment could result in less toxicity. Multiple studies have evaluated potential ways to de-escalate treatment and reduce toxicity, such as dose reduction or change of chemotherapeutic agent. Another possible de-escalation strategy, which is pursued here, is to reduce the elective clinical target volume.

A multi-institutional dataset of 598 oropharyngeal SCC patients in whom the detailed patterns of lymph node involvement are reported was collected. The publicly available online platform www.LyProX.org was developed to share and visualize the data. Based on this data, a statistical model of lymphatic tumor progression to perform a statistical analysis to estimate the probability of occult metastases in the clinically negative lymph node levels was developed. The patient's state of metastatic lymphatic progression is described via a hidden Markov model. The state of tumor progression is described by a collection of hidden binary random variables that indicate the involvement of lymph node levels. The model parameters are the probabilities for the tumor to spread to and between lymph node levels and are learned from the dataset. Supporting clinical experience, these statistical calculations can subsequently be used as a basis, to personalize the risk estimation of occult lymph node metastases in newly diagnosed patients based on their distribution of macroscopic metastases, T-stage, and lateralization of the primary tumor. A table with the possible different combinations of clinically observed lymph node involvement and the associated risk of occult lymph node involvement in the remaining, clinically negative lymph node levels (LNL) was created. By interpreting the results from both the statistical analysis and clinical experience, the elective clinical target volume (CTV) was personalized based on a patient's individualized risk profile. As a final measure of quality assurance, the elective CTVs (CTV-3s) constructed in this way have been discussed individually by the investigators, to ensure consistency with data and clinical judgement and experience. This leads to a reduction of irradiated volume and, potentially, to a reduction in early and late toxicity.

The aim of this clinical trial is to determine the safety of the use of a personalized de-escalated elective nodal CTV in oropharynx SCC patients treated with primary (chemo)radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a newly diagnosed (no pre-treatment) squamous cell carcinoma of the oropharynx (i.e. tonsils, base of tongue, oropharyngeal walls, oropharyngeal surface of epiglottis; ICD-10 codes C01, C09, C10), T1-4, N0-3.
* Treatment with definitive (chemo) radiotherapy planned, with elective irradiation of the lymph nodes.
* Age ≥ 18 years, no upper age limit.
* ECOG performance score < 3.
* History/physical examination within 30 days prior to study inclusion by head and neck surgeon and/or radiation oncologist.
* FDG-PET scan prior to study inclusion. In case of inability to perform or contra-indication, at least contrast enhanced MRI scan obligatory.
* Participants need to provide informed consent.

Exclusion Criteria:

Inclusion Criteria:

* Patients with a newly diagnosed (no pre-treatment) squamous cell carcinoma of the oropharynx (i.e. tonsils, base of tongue, oropharyngeal walls, oropharyngeal surface of epiglottis; ICD-10 codes C01, C09, C10), T1-4, N0-3.
* Treatment with definitive (chemo) radiotherapy planned, with elective irradiation of the lymph nodes.
* Age ≥ 18 years, no upper age limit.
* ECOG performance score < 3.
* History/physical examination within 30 days prior to study inclusion by head and neck surgeon and/or radiation oncologist.
* FDG-PET scan prior to study inclusion. In case of inability to perform or contra-indication, at least contrast enhanced MRI scan obligatory.
* Participants need to provide informed consent.

Exclusion Criteria:

* Multilevel primary tumors extending unambiguously beyond the oropharynx into the oral cavity, naso- or hypopharynx
* Distant metastases detected.
* Previous surgery, chemotherapy or radiotherapy treatment for other head and neck cancers.
* Previous surgery in head and neck region affecting the cervical lymphatic system. Dissection of singular lymph nodes for diagnostic purposes before treatment start is allowed.
* Synchronous or previous malignancies. Exceptions are curatively treated basal cell carcinoma or SCC of the skin, or in situ carcinoma of the cervix uteri, low- or intermediate- risk prostate cancer or breast with a progression-free follow-up time of at least 3 years without any remaining disease burden, or other previous malignancy with a progression-free interval of at least 5 years without any remaining active/progressive disease burden regardless whether the treatment is completed or ongoing as a maintenance treatment (e.g. androgen deprivation therapy for prostate cancer).
* Pregnancy or breast feeding
* Any severe mental or psychic disorder affecting decision making and ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
out-of field nodal recurrence rate at 2 years | from completion of treatment up to 2 years after radiotherapy
  efficacy of personalized CTV-N reduction in oropharyngeal SCC patients 2 years after the end of the primary (chemo)radiotherapy treatment measured by the Kaplan-Meier estimator for the cumulative probability of out-of-field N-site recurrences (incidence of lymph node metastases in non-irradiated LNLs).

SECONDARY OUTCOMES:
out-of field nodal recurrence rate at 3 years | from completion of treatment up to 3 years after radiotherapy
  efficacy of personalized CTV-N reduction in oropharyngeal SCC patients measured by the Kaplan-Meier estimator for the cumulative probability of out-of-field N-site recurrences (incidence of lymph node metastases in non-irradiated LNLs)
Loco-regional control (LCR) rate at 2 years | from completion of treatment up to 2 years after radiotherapy
  assessed by the Kaplan-Meier estimator for the cumulative probability of local recurrence of the primary tumor or recurrence in any cervical LNL (both irradiated and non-irradiated LNLs)
Loco-regional control (LCR) rate at 3 years | from completion of treatment up to 3 years after radiotherapy
  assessed by the Kaplan-Meier estimator for the cumulative probability of local recurrence of the primary tumor or recurrence in any cervical LNL (both irradiated and non-irradiated LNLs)
Progression-free survival (PFS) at 2 years | from completion of treatment up to 2 years after radiotherapy
  assessed by the Kaplan-Meier estimator for the cumulative probability of any local, regional, distant progression or death
Progression-free survival (PFS) at 3 years | from completion of treatment up to 3 years after radiotherapy
  assessed by the Kaplan-Meier estimator for the cumulative probability of any local, regional, distant progression or death
Overall Survival (OS) at 2 years | from completion of treatment up to 2 years after radiotherapy
  assessed by the Kaplan-Meier estimator for the cumulative probability of death from any cause
Overall Survival (OS) at 3 years | from completion of treatment up to 3 years after radiotherapy
  assessed by the Kaplan-Meier estimator for the cumulative probability of death from any cause
Early toxicity of treatment | treatment start up to 3 months after treatment
  assessed by grading of toxicities according to CTCAE v5.0 - overall toxicity will be evaluated according to the TAME methodology.
Late toxicity of treatment | >3 months up to 3 years after treatment
  assessed by grading of toxicities according to CTCAE v5.0 - overall toxicity will be evaluated according to the TAME methodology.
Overall Quality of life at end of treatment | at the last day of radiotherapy (+/- 1week)
  assessed according to paper-based questionnaires EORTC QLQ C30 All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems
Quality of life regarding head and neck specific symptoms at end of treatment | at the last day of radiotherapy (+/- 1week)
  assessed according to paper-based questionnaires, i.e. head and neck module HN43: All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems
Overall Quality of life at 6 months after treatment | at 6 months after the last day of radiotherapy (+/- 2 weeks)
  assessed according to paper-based questionnaires EORTC QLQ C30: All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems
Quality of life regarding head and neck specific symptoms at 6 months after treatment | at 6 months after the last day of radiotherapy (+/- 2 weeks)
  assessed according to paper-based questionnaires, i.e. head and neck module HN43: All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems
Overall Quality of life at 12 months after treatment | at 12 months after the last day of radiotherapy (+/- 2 weeks)
  assessed according to paper-based questionnaires EORTC QLQ C30: All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems
Quality of life regarding head and neck specific symptoms at 12 months after treatment | at 12 months after the last day of radiotherapy (+/- 2 weeks)
  assessed according to paper-based questionnaires, i.e. head and neck module HN43: All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems
Overall Quality of life at 24 months after treatment | at 24 months after the last day of radiotherapy (+/- 2 weeks)
  assessed according to paper-based questionnaires EORTC QLQ C30: All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems
Quality of life regarding head and neck specific symptoms at 24 months after treatment | at 24 months after the last day of radiotherapy (+/- 2 weeks)
  assessed according to paper-based questionnaires, i.e. head and neck module HN43: All of the scales and single-item measures range in score from 0 to 100. A high scale score A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems

OTHER OUTCOMES:
Assessement of values and longitudinal changes in total blood count, including lymphocytes (explorative assessement) | Treatment start and every 3 months up to 3 years after radiotherapy
  Full blood count will be longitudinally assessed at begin of treatment and at every follow up (descriptive analyses and correlation with all oncological outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Balermpas, MD, Principal Investigator — University of Zurich
Locations (5):
- Switzerland (5):
  - Zurich University Hospital, Zurich, Canton of Zurich
  - Cantonal Hospital Aarau, Aarau
  - Ospedale Regionale di Bellinzona, Bellinzona
  - Inselspital Bern, Bern
  - Hôpitaux universitaires de Genève, Geneva

IPD SHARING:
Plan to Share IPD: No